CLINICAL TRIAL: NCT00517699
Title: An Open Label Study of the Effect of Rituxan, High Dose Methotrexate and High Dose Cytarabine on Response Rate in Patients With Primary Central Nervous System Lymphoma.
Brief Title: A Study of MabThera (Rituximab) in Primary Central Nervous System Lymphoma.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early due to lack of enrollment.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML19652
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Results first posted 2014-08-08 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-07

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Rituximab; Methotrexate; Cytarabine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: Methotrexate; Drug: Cytarabine

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 750mg/m2 iv
Drug: Methotrexate — 8g/m2 iv
Drug: Cytarabine — 2g/m2 iv

SUMMARY:
This study will evaluate the efficacy and safety of MabThera plus high dose methotrexate plus high dose cytarabine in patients with central nervous system non-Hodgkin's lymphoma. Eligible patients will receive a treatment regimen consisting of MabThera (750mg/m2 iv) plus methotrexate (8g/m2 iv) given at intervals up to week 22, plus cytarabine (2g/m2 iv) at week 11 and week 22. The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-80 years of age;
* histological diagnosis of primary central nervous system lymphoma;
* B-cell proliferation verified by positive staining for CD20;
* >=1 measurable lesion.

Exclusion Criteria:

* prior chemotherapy, other than corticosteroids, >=6 weeks before and after diagnosis or surgery;
* history of prior cranial irradiation;
* evidence of plurisystemic non-Hodgkin's lymphoma;
* other active malignant disease (other than basal cell or squamous cell cancer of skin,or cancer in situ of cervix;
* uncontrolled active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Canada (2):
  - Greenfield Park, Quebec
  - Québec, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab, Cytarabine, and Methotrexate (MTX): Participants received single doses of rituximab 750 milligrams per square meter (mg/m^2) intravenously (IV) at Weeks 1 through 5, and 7, 9, 11, 14, 16, 18, 20, and 22; cytarabine 2 grams per square meter (g/m^2) IV every 24 hours for 2 doses at Weeks 11 and 22; and single doses of MTX 8 g/m^2 IV at Weeks 3, 5, 7, 9, 14, 16, 18, and 20.
Period: Overall Study
Arm/Group | Rituximab, Cytarabine, and Methotrexate (MTX)
Started | 5
Completed | 0
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1
Not completed — Administrative error | 1
Not completed — Study terminated by Sponsor | 2

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received any amount of study drug.
Groups:
- Rituximab, Cytarabine, and MTX: Participants received single doses of rituximab 750 mg/m^2 IV at Weeks 1 through 5, and 7, 9, 11, 14, 16, 18, 20, and 22; cytarabine 2 g/m^2 IV every 24 hours for 2 doses at Weeks 11 and 22; and single doses of MTX 8 g/m^2 IV at Weeks 3, 5, 7, 9, 14, 16, 18, and 20.
Arm/Group | Rituximab, Cytarabine, and MTX
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (8.23) [47 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Complete Response (CR) or Unconfirmed CR (CRu)
Description: CR: complete disappearance of all enhancing abnormalities on contrast-enhanced cranial magnetic resonance imaging (MRI); no evidence of active ocular lymphoma as defined by absence of cells in the vitreous and resolution of any previously documented retinal or optic nerve infiltrates; negative cerebrospinal fluid (CSF) cytology; at the time of CR determination, participant had discontinued use of all corticosteroids for at least 2 weeks. CRu requires fulfillment of CR criteria but with these limitations: Fulfills CR criteria but had continued requirement for corticosteroid therapy at any dose; small but persistent enhancing abnormality on MRI related to biopsy or focal hemorrhage; persistent minor abnormality on follow-up ophthalmologic exam (related to persistent non-malignant cells in vitreous, or alterations in retina/optic nerve not consistent with tumor infiltration) if the abnormality is unlikely to represent ocular lymphoma.
Time Frame: Week 24
Population: Due to early study termination, all efficacy data were documented by data listings only, no data analysis was performed.
Arm/Group | Rituximab, Cytarabine, and MTX
Number analyzed (Participants) | 0

2. Primary Outcome: Percentage of Participants With a CR, CRu or Partial Response (PR)
Description: PR: greater than or equal to (≥) 50 percent (%) decrease in the contrast-enhancing lesion seen on MRI as compared with the baseline images; (2) Corticosteroid dose was irrelevant to the determination of PR; for participants with ocular disease, ophthalmologic exam must show a decrease in vitreous cell count or retina/optic nerve cellular infiltrate but may have continued to show persistent malignant or suspicious cells; for participants with CSF positive for neoplastic cells, CSF cytology may be negative or continue to show persistent malignant or suspicious cells in patients with ≥50% decrease in the primary brain lesions; no new sites of disease.
Time Frame: Week 24
Population: Due to early study termination, all efficacy data were documented by data listings only, no data analysis was performed.
Arm/Group | Rituximab, Cytarabine, and MTX
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants With Initial CR or CRu and Subsequent Disease Relapse
Time Frame: Week 24
Population: Due to early study termination, all efficacy data were documented by data listings only, no data analysis was performed.
Arm/Group | Rituximab, Cytarabine, and MTX
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: Time from entry into trial until death of any cause. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last dose and participants with no post baseline information were censored at the baseline date.
Time Frame: Time of last follow-up assessment between Day 1 and 3 years
Population: Due to early study termination, all efficacy data were documented by data listings only, no data analysis was performed.
Arm/Group | Rituximab, Cytarabine, and MTX
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time interval between the entry into trial and occurrence of one of the following events: progression of disease (PD) or death as a result of primary central nervous system lymphoma (PCNSL). Participants who were withdrawn from the study without documented progression and for whom there existed case report form (CRF) evidence that evaluations had been made, were censored at the date of last tumor assessment when participant was known to be progression free. Participants without postbaseline tumor assessments but known to be alive were censored at the time of randomization. PD required a ≥25% increase in the contrast-enhanced lesion seen on MRI as compared with baseline or best response (comparison should be made to the smallest of multiple lesions); progression of ocular disease as indicated by an increase in vitreous cell count or progressive retinal or optic nerve infiltration, appearance of any new lesion or site of disease during or at the end of therapy.
Time Frame: Week 24
Population: Due to early study termination, all efficacy data were documented by data listings only, no data analysis was performed.
Arm/Group | Rituximab, Cytarabine, and MTX
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 24 weeks.
Arm/Group | Rituximab, Cytarabine, and MTX
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab, Cytarabine, and MTX (N=5)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Eye allergy (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 3
Generalised oedema (General disorders) | 2
Hyperthermia (General disorders) | 3
Injection site erythema (General disorders) | 1
Injection site pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 1
Vessel puncture site bruise (General disorders) | 1
Hepatitis (Hepatobiliary disorders) | 1
Conjunctivitis bacterial (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Drug toxicity (Injury, poisoning and procedural complications) | 3
Skin laceration (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Creatinine renal clearance decreased (Investigations) | 1
Hepatic enzyme abnormal (Investigations) | 1
Hepatic enzyme increased (Investigations) | 2
Weight increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5
Malnutrition (Metabolism and nutrition disorders) | 1
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Dementia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Loss of consciousness (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusional state (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Arterial thrombosis limb (Vascular disorders) | 1
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.